CLINICAL TRIAL: NCT04146233
Title: An Observer Blinded Point-of-care Gastric Ultrasound Analysis of the Gastric Emptying Time of Orange Juice With and Without Pulp
Brief Title: POCUS Analysis of the Gastric Emptying Time of Orange Juice With and Without Pulp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Christopher Wahal, Assistant Professor of Anesthesiology, Thomas Jefferson University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19D.577
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Preoperative Period; Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Ultrasound images will be saved and reviewed by blinded investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange Juice without pulp (Other): Drink orange juice without pulp and have gastric ultrasound performed 2 hours later
  Interventions: Other: Point of care gastric ultrasound
- Orange juice with pulp (Other): Drink orange juice with pulp and have gastric ultrasound performed 2 hours later
  Interventions: Other: Point of care gastric ultrasound

INTERVENTIONS:
Other: Point of care gastric ultrasound — Point-of-care gastric ultrasound will be performed using a low-frequency curvilinear ultrasound probe to assess stomach contents (empty vs. not empty, liquid vs. solid, gastric volume).

SUMMARY:
Preoperative fasting guidelines for anesthesia recommend waiting two hours after ingesting a clear liquid and six hours after ingesting a light meal. Due to the presence of pulp, orange juice is considered a light meal by current guidelines which means a patient must wait six hours before undergoing general anesthesia. This study will use ultrasound of stomach of healthy volunteers to determine if the presence of pulp actually increases the transit time for orange juice.

DETAILED DESCRIPTION:
Healthy volunteers will be solicited (medical students and attending anesthesiologists) to participate in the study. Volunteers will participate in two sessions, one for orange juice without pulp and one for orange juice with pulp. Participants will be NPO after midnight and will be asked to arrive at approximately 8 am. Upon arrival for females of child bearing age, a urine pregnancy test will be performed and they will be discreetly informed of the results of the test. After, all patients will have their gastric volume assessed using point-of-care ultrasound to ensure the study team is able to adequately identify their stomach as well as to ensure the stomach is empty. After measurements are made, participants will drink 12 oz (approximately 350 mL) of either orange juice with or without pulp. Two hours after finishing the juice they will again undergo point-of-care gastric ultrasound scanning. Images will be saved and will be examined by a blinded independent anesthesiologist. The study will entail two visits each lasting for approximately 3 hours.

Point-of-care gastric ultrasound will be performed using a low-frequency curvilinear ultrasound probe. The exam will be performed on a stretcher with the participant in both the supine and right lateral decubitus (RLD) position. The goal of point-of-care gastric ultrasound is to obtain an image of the gastric antrum. The low-frequency large curvilinear probe is placed in the epigastric area in a sagittal or parasagittal plane immediately inferior to the patient's xiphisternum with the orientation marker directed cephalad. Image optimization requires scanning in an anterior and cephalad direction toward the liver by tilting the tail of the probe toward the feet. A qualitative analysis will occur first to rule out solid contents in the stomach. Once confirmed, the gastric antral cross-sectional area (CSA) will be measured in the RLD position. Correlation has been shown between CSA and total gastric fluid volume. A gastric volume less than 1.5 mL/kg is considered consistent with fasting.

The study will be repeated for both orange juice with and without pulp.

ELIGIBILITY:
Inclusion Criteria:

* volunteers age 18-65 years old, American Society of Anesthesiologists physical status 1-2

Exclusion Criteria:

* presence of diabetes mellitus, previous gastric surgery, presence of hiatal hernia, history of delayed gastric emptying, pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Assessment of Gastric Volume at 2 hours | 2 hours after intervention
  Two hours after orange juice (with and without pulp) is consumed, point of care gastric ultrasound will be used to assess gastric contents and gastric volume

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wahal, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No